CLINICAL TRIAL: NCT07177846
Title: LiveWell: An Adapted Dialectical Behavioral Therapy Skills Training Protocol for Patients Living With Metastatic Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kelly Hyland, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00144605; R00CA286959 (NIH)
Record Dates: First submitted 2025-09-08; First posted 2025-09-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Survivorship
Keywords: Dialectical Behavioral Therapy; Psychosocial Oncology; Lung Cancer; Psychological Distress
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LiveWell: An Adapted Dialectical Behavioral Therapy Skills Training Program (Experimental): Will receive 8 telehealth sessions delivered 1 on 1 via telehealth with a trained mental health professional. Sessions will be delivered approximately weekly and are 45-60 min in length. Sessions will teach skills from dialectical behavioral therapy (e.g., mindfulness, distress tolerance, emotion regulation, interpersonal effectiveness) adapted for patients with metastatic lung cancer. Sessions follow a standardized structure, including 1) mindfulness practice, 2) home practice and diary card review, 3) learning and practicing new skills, and 4) closing ritual. Participants will have access to a resource library of skills training videos and mindfulness recordings.
  Interventions: Behavioral: LiveWell: An Adapted Dialectical Behavioral Therapy Skills Training Program
- Usual Care (No Intervention): Will receive a handout with general support resources available at Hollings Cancer Center.

INTERVENTIONS:
Behavioral: LiveWell: An Adapted Dialectical Behavioral Therapy Skills Training Program — LiveWell: Adapted DBT Skills Training for Patients with Metastatic Lung Cancer
  Arms: LiveWell: An Adapted Dialectical Behavioral Therapy Skills Training Program

SUMMARY:
In this pilot randomized controlled trial, patients with metastatic non-small cell lung cancer and at least mild distress (N=80) will be randomized to receive LiveWell, an adapted Dialectical Behavioral Therapy (DBT) Skills Training protocol) or Usual Care. The investigators will evaluate feasibility, acceptability, and preliminary efficacy of LiveWell to reduce distress (primary outcome) and improve psychological well-being, symptom burden, and quality of life (secondary outcomes). The investigators will explore emotion regulation as a potential mechanism of change.

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to receive LiveWell, an eight-session, telehealth-delivered DBT Skills Training intervention tailored for lung cancer metavivors, or Usual Care. Participants will complete self-report measures at baseline, 8-week follow-up, and 3 month follow-up. It is hypothesized that: 1) RCT methods will demonstrate evidence of feasibility (accrual N=80/20 months, >80% adherence to assigned interventions and assessments, <25% attrition) and acceptability (>3/5 satisfaction study procedures, >3 mean intervention satisfaction LiveWell); 2) LiveWell participants will demonstrate reductions in distress (primary outcome) and improvements in psychological well-being (illness acceptance, positive affect, tolerance of uncertainty, mindfulness, self-efficacy to manage emotions and symptoms), symptom burden (fatigue, dyspnea, pain), and quality of life (secondary outcomes) compared to Usual Care participants at 8-week follow-up. H3. (Exploratory). To explore the role of emotion regulation as a potential mechanism of change.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* AJCC Stage IV non-small cell lung cancer
* Receiving treatment with non-curative intent
* English proficiency
* Able to provide informed consent
* National Comprehensive Cancer Network distress screening score ≥ 3/10

Exclusion Criteria:

* Cognitive impairment
* Untreated serious mental illness
* Expected survival < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
PROMIS Anxiety Short Form (8a) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  Anxiety will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety (8 items) Short Form Scale. PROMIS scores are expressed as T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate greater anxiety symptomology.
PROMIS Depression Short Form (8a) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  Depression will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (8 items) Short Form Scale. PROMIS scores are expressed as T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate greater depressive symptomology.

SECONDARY OUTCOMES:
Intolerance of Uncertainty Scale - Short Form (IUS-12) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The 12-item Intolerance of Uncertainty Scale (IUS) Short Form will be used to measure emotional, cognitive, and behavioral reactions to uncertain situations. The IUS has a score range of 12-60, where a higher score indicates greater intolerance of uncertainty.
Peace, Equanimity, and Acceptance in the Cancer (PEACE) - Peaceful Acceptance of Illness Subscale | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The 5-item Peace, Equanimity, and Acceptance in the Cancer (PEACE) - Peaceful Acceptance of Illness Subscale will be used to assess patient-reported acceptance, inner peace, and tranquility in the context of cancer. The subscale has a score range of 5-20, where a higher score indicates greater peaceful acceptance of illness.
PROMIS Positive Affect Short Form (15a) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The PROMIS Positive Affect Short Form 15a will be used to assess patient-reported positive emotions and well-being over the past 7 days. PROMIS scores are expressed as T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate greater positive affect.
Difficulty in Regulating Emotions Scale (DERS-18) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The DERS-18 will be used to assess emotion dysregulation. The DERS-18 has a score range of 18-80, where a higher score indicates greater difficulty with regulating emotions.
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The 10-item Cognitive and Affective Mindfulness Scale-Revised will be used to assess patient-reported mindfulness qualities, including present-moment awareness, acceptance, and attention. The CAMS-R has a score range of 10-40, where a higher score indicates greater mindfulness.
PROMIS Self-Efficacy for Managing Symptoms Short Form (8a) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The PROMIS Self-Efficacy for Managing Symptoms 8-item Short Form will be used to assess patient-reported confidence in managing symptoms and limiting their interference with daily life. PROMIS scores are expressed as T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate greater self-efficacy for managing symptoms.
PROMIS Self-Efficacy for Managing Emotions (8a) Short Form | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  PROMIS Self-Efficacy for Managing Emotions 8-item Short Form will be used to assess patient-reported confidence in managing negative emotions and emotional distress related to chronic illness. PROMIS scores are expressed as T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate greater self-efficacy for managing emotions.
NCI Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (NCI-PRO-CTCAE) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The NCI-PRO-CTCAE will be used to assess patient-reported symptom frequency, severity, and interference related to lung cancer and its treatment. Items are rated on a 5-point Likert scale, with higher scores indicating greater symptom burden.
Functional Assessment of Cancer Therapy - Lung (FACT-L) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The FACT-L will be used to assess patient-reported quality of life across physical, social/family, emotional, and functional domains, as well as lung cancer-specific concerns. Items are rated on a 5-point Likert scale (0 = Not at all to 4 = Very much) and summed to form subscale and total scores. Higher subscale and total scores indicate better quality of life.
DBT Ways of Coping Checklist (DBT-WCCL) - DBT Skills Subscale (DSS) | Baseline (week 0), post-intervention (week 8), and 3 month follow-up (week 20)
  The DBT Ways of Coping Checklist (DBT-WCCL) -DBT Skills Subscale (DSS) will be used to assess patient-reported frequency of skill use to manage difficult situations. The DBT-WCCL has a score range of 0 to 4, where a higher score indicates greater DBT skill use.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Hyland, PhD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Final datasets for analyses will include outcome measures and any derived variables necessary to answer the Specific Aims along with demographic characteristics. Raw data will be collected via self-report survey links from the research participants and stored in the REDCap research database. Data will be exported to SAS for data cleaning and derivation of outcome variables, as necessary. Any changes to the raw data will be corrected directly in REDCap while logging reasons for the edits. All datasets that can be shared will be deposited in the NIMH Data Archive (NDA; https://nda.nih.gov), a publicly maintained data archive whose mission is to accelerate scientific research and discovery through data sharing, data harmonization, and the reporting of research results. The NDA provides metadata, persistent identifiers, and long-term access. This repository is supported by the NIH. The PI, Dr. Hyland, will be responsible for ensuring compliance with the data management sharing plan.
Supporting Information: Study Protocol
Time Frame: Shared data for this study will be shared with the NDA and available for request no later than at time of publication of primary results or the end of performance period, whichever comes first. The shared data deposited in the NDA will exist indefinitely.
Access Criteria: Data deposited to the NDA will exist indefinitely and may be accessed by any individual in alignment with the terms set forth by NIH on this NIH-sponsored data repository site (https://nda.nih.gov/nda/access-datainfo), as well as privacy and confidentiality protections such as the NIH Certificate of Confidentiality and applicable laws, regulations, and policies governing data derived from human participants. Access to scientific data will be controlled via safeguards and protections currently in place via the NDA. To ensure participant consent for data sharing, IRB paperwork and informed consent documents will include language describing plans for data management and sharing data, describing the motivation for sharing, and explaining that personal identifying information will be removed. To protect participant privacy and confidentiality, shared data will be de-identified by stripping all PHI data and including the GUID to link all research data.